CLINICAL TRIAL: NCT03528486
Title: Interventions to Attenuate Cognitive Decline
Brief Title: Interventions to Attenuate Cognitive Decline: Keys to Staying Sharp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Jerri D. Edwards, Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 32335
Record Dates: First submitted 2018-03-13; First posted 2018-05-17 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Age-related Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Training I (Experimental): Participants will complete a type of music training including listening to music, learning about music, or learning to read music, or play a musical instrument.
  Interventions: Behavioral: Music Training I
- Music Training II (Active Comparator): Participants will complete a type of music training including listening to music, learning about music, or learning to read music, or play a musical instrument
  Interventions: Behavioral: Music Training I

INTERVENTIONS:
Behavioral: Music Training I — Participants will be attending group classes, guided by a trainer, with up to 10 other older adults.

SUMMARY:
Different cognitive intervention approaches have been developed to attenuate decline (e.g., cognitive engagement, training, or stimulation), but it is not clear which approaches are efficacious. It is also not clear when, along the continuum of normal cognitive aging to mild cognitive impairment (MCI-a transitional stage before dementia onset), it is most efficacious to intervene. This randomized clinical trial will determine the efficacy of a novel cognitive engagement intervention approach (music training) as compared to cognitive stimulation (which will serve as a stringent, active control). Grounded in theory, the central hypothesis is that interventions enhancing central auditory processing (CAP), a strong, longitudinal predictor of MCI and dementia, will improve cognition. Music training is increasingly recognized as a feasible means to attenuate age-related cognitive decline. Prior research and preliminary data suggest that intense piano training enhances CAP and is likely more effective than cognitive stimulation. Correlational studies indicate superior CAP, executive function, and other cognitive abilities for adults with formal music training compared to non-musicians. The specific aims of the study are to examine the efficacy of music training relative to cognitive stimulation (active controls) to improve CAP, cognition, and everyday function among older adults with and without MCI. The efficacy of music training will be established and moderating effects of MCI status will be examined. The proposed study further aims to elucidate the underlying mechanisms of effective cognitive intervention approaches by exploring mediators of training gains. The proposed study is the first phase II randomized trial of music training to enhance older adults' cognition. Mediation analyses will elucidate the underlying mechanisms of intervention effects.

DETAILED DESCRIPTION:
Interventions to Attenuate Cognitive Decline: Keys to Staying Sharp.

The primary objectives is to examine the efficacy of music training to improve central auditory processing (CAP), cognition, and everyday function among older adults.

The secondary objectives are:

* To examine the moderating effects of mild cognitive impairment (MCI) on music training efficacy.
* To explore mediators of intervention effects.

Design The design is a two arm randomized clinical trial examining the efficacy of music training to improve CAP, cognition, and everyday function in older adults with and without MCI across two time points (baseline and immediate post-test).

Outcomes The effects of of music training on CAP, cognition, and everyday functional performance will be quantified.

CAP processing measures will include: Time Compressed Speech 65%, Words-in-Noise, Dichotic Digits Test, Dichotic Sentence Identification, and Adaptive Tests of Temporal Resolution. A composite will be derived from principal components analyses.

Cognition measures will include: Verbal Fluency Test (phonemic fluency, category fluency, and category switching), Trail Making Test, and Digit Coding. A composite will be derived from principal component analyses.

Everyday Function measures will include: Timed Instrumental Activities of Daily Living and Test of Everyday Attention. A composite will be derived from principal component analyses.

Interventions and Duration Two types of music training will be investigated. The two training conditions will be equivalent in terms of frequency and duration of each session (90 min/day, two days/wk, 10 weeks) and social contact (led by trainer and conducted in groups of up to 10 persons).

Sample Size and Population In-person screening of a maximum of 500 potential study participants are planned to enroll up to 400 participants. The goal is to have at least 200 participants complete the study. Individuals with normal cognition and those with a clinical diagnosis of MCI will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or older
* willingness to provide informed consent
* willingness to complete up to 23 study visits including attending in-lab intervention two times a week for a three-month period with the goal of completing 20 sessions.
* ability to speak and understand English
* Montreal Cognitive Assessment score of 20 or higher (score 20 to 30 inclusive)
* intact vision (binocular near visual acuity of 20/50 or better tested with a standard near visual acuity chart)
* adequate hearing acuity (no greater than a moderate hearing loss [thresholds <70 dB HL] in the mid-frequency range [1000, 2000 Hz] in at least one ear as determined by a standard pure tone hearing evaluation)
* Music Reading Assessment score of 18 or lower (score 0-18 inclusive)
* ability to understand study procedures and comply with them for the length of the study in the tester's opinion (and other study personnel opinion who interact with participant, such as the study physician)

Exclusion Criteria:

* moderate or worse depressive symptoms (Geriatric Depression Scale short form score >=5)
* previous participation in University of South Florida (USF) Cognitive Aging Lab intervention studies
* previous participation in 10 or more hours of a computerized cognitive intervention computer programs (e.g., Lumosity, Posit Science Brain Fitness, InSight, or BrainHQ; Lace, CogMed, CogniFit, Happy Neuron, Dakim, DriveSharp or Staying Sharp programs)
* currently enrolled in another research study
* planning on being away for two or more weeks during the next five months (recruit later)
* undergoing chemotherapy or radiation treatment or planning surgeries or other procedures requiring anesthesia within the next five months (recruit later)
* four or more years of formal music training such as private lessons or group lessons on a specific instrument
* ability to read music on two or more of the following clefs: Treble clef, Bass clef, Alto clef
* four or more years of playing any one musical instrument
* currently practicing or participating in any music activities- such as music performance or music reading or music lessons
* difficulty and pain in moving hands or fingers, or neuropathy affecting hands, or tremor in either hand
* self-reported diagnosis of dementia, stroke, serious brain injury or neurological disorder
* diagnosed by a physician or nurse with a TIA that occurred within the last 18 months
* inability or unwillingness to give written informed consent at baseline
* Clinical Dementia Rating Scale score of 1 or greater
* Clinical diagnosis of dementia or other disorder that in the study physician's opinion would limit the persons ability to participate in the study or benefit from the interventions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Cognition | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  A composite of performance on Verbal fluency words generated, Trail Making Test time, and Digit Symbol Coding number correct derived from principal components analyses

SECONDARY OUTCOMES:
Central Auditory Processing | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  A composite will be formed from principal components analyses of number correct for performance on Time Compressed Speech Test (TCS), Words-in-Noise Test (WIN), Dichotic Digits Test (DDT), Dichotic Sentence Identification (DSI) and the threshold in ms of performance on the Adaptive Tests of Temporal Resolution (ATTR).
Everyday Function | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  A composite will be formed from the time and accuracy of performance on the Timed IADL Test and The Test of Everyday Attention (TEA)

OTHER OUTCOMES:
General Self Efficacy | Change from prior to training content exercises to immediately after training content exercises, at the end of intervention phase which is about three months
  General Self-Efficacy scale likert scaling with higher numbers reflecting better self efficacy. 23 items on a 14-point scale. Items will be summed. Items are designed to reflect effort, initiation, and persistence as described by Bandura
Music Self Efficacy | Change from prior to training content exercises to immediately after training content exercises, at the end of intervention phase which is about three months
  Music Self-Efficacy scale likert scaling with higher numbers reflecting better music self efficacy. 24 items with liker scaling of 1 to 100. Total across all items will be summed. Items reflect the degree to which participants have positive feelings and beliefs in their musical abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Runge SK, Hudak EM, Sutfin JA, Dobrovolskiy VR, Edwards JD. The influence of peer navigators on intervention adherence and retention among older adults: A study within a randomized trial - SWAT. Contemp Clin Trials. 2025 Dec 24;161:108206. doi: 10.1016/j.cct.2025.108206. Online ahead of print. PMID 41453521
- [Derived] Hudak EM, Bugos J, Andel R, Lister JJ, Ji M, Edwards JD. Keys to staying sharp: A randomized clinical trial of piano training among older adults with and without mild cognitive impairment. Contemp Clin Trials. 2019 Sep;84:105789. doi: 10.1016/j.cct.2019.06.003. Epub 2019 Jun 18. PMID 31226405

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03528486/Prot_SAP_001.pdf